CLINICAL TRIAL: NCT02400619
Title: Efficacy of Radial Extracorporeal Shock Waves Compared to Botulinum Toxin Type A in the Treatment of Spasticity of the Lower Extremities in Patients With Cerebral Palsy: a Crossover Randomized Clinical Trial.
Brief Title: Shockwaves Therapy and Botulinum Toxin for the Treatment of Spasticity in Patients With Cerebral Palsy. A Cross Over RCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Xavi Vidal Novellas (Other)
Collaborators: Cerebral Palsy Association (Other)
Responsible Party: Sponsor-Investigator, Xavi Vidal Novellas, Xavi Vidal Novellas Health Sciences Faculty Blanquerna and physical therapist in Aspace Association of Cerebral Palsy, University Ramon Llull
Organization: University Ramon Llull (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: Neuroshockwaves
Record Dates: First submitted 2015-03-06; First posted 2015-03-27 (Estimated); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Spasticity; Cerebral Palsy
Keywords: shockwaves; Physiotherapy; Botulinum toxin
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- shock waves (Active Comparator): A comparative study with patients with spasticity in gastrocnemius and soleus where a group start having shockwave treatment and receive three sessions at weekly intervals, gastrocnemius and soleus applied in 2000 impacts at a frequency of 8hz and energy intensity is proposed between 2.2-2.4 Bars (0,10-0,12mj ). Swiss dolor clast EMS. The other group will receive botulinum toxin Type A in the same muscles. The dose of toxin is in accordance with the weight of each patient, the dose normally used with each user and always with the same brand is always respected, Botox (4-8-12 U/Kg) Patients will be assessed before treatment, after three weeks, two months and three months after three months when the groups exchange the therapy.
  Interventions: Device: shock waves
- botulinum toxin (Active Comparator): A comparative study with patients with spasticity in gastrocnemius and soleus where a group start having shockwave treatment and receive three sessions at weekly intervals, gastrocnemius and soleus applied in 2000 impacts at a frequency of 8hz and energy intensity is proposed between 2.2-2.4 Bars (0,10-0,12mj ). Swiss dolor clast EMS.The other group will receive botulinum toxin type A in the same muscles. The dose of toxin is in accordance with the weight of each patient, the dose normally used with each user and always with the same brand is always respected. Botox (4-8-12 U/Kg)Patients will be assessed before treatment, after three weeks, two months and three months after three months when the groups exchange the therapy.
  Interventions: Drug: Botulinum Toxin Type A

INTERVENTIONS:
Device: shock waves — Swiss dolorclast smart EMS Registration: EN-60601-1 Type BF IP40. 93/42 CEE
  Arms: shock waves
Drug: Botulinum Toxin Type A — Botulinum toxin type A Botox
  Other Names: Type A
  Arms: botulinum toxin

SUMMARY:
Spasticity is a motor disorder that can affect the lower limbs in up to 75% patients with cerebral palsy, having a significantly effect on their mobility and quality of life. There is much controversy about what is the most appropriate treatment of spasticity The objective of the present study is to evaluate the effects of radial extracorporeal shock wave therapy (rESWT) compared to treatment with botulinum toxin to improve spasticity in patients with cerebral palsy

The number needed of patients is 70 (35 per group). Leaving a period of washout between one therapy and the other

DETAILED DESCRIPTION:
Outcome Measures:

The primary outcome will be to measure spasticity with passive range of motion of the foot (pROM) by muscular extensibility and its traction reflex using goniometryIt will be assessed at baseline before the treatment, as well as after 3 weeks, 2 months, 3 months, after the washout period (3months), 3 months and 3 weeks, 5 months and 6 months, when the end the intervention.

Secondary outcome includes: 1) Pain will be assessed with Visual Analog Scale (VAS) after the first application of each therapy. 2) Ascertain if the type of Gross Motor Functional Classification System (GMFCS) has an influence on the improvement of these two treatments; 3) Assess whether infiltration of Botulinum Toxin in other muscle groups have influence on the results of study; and 4) Undergo a qualitative registration to know the perception and experience that patient/family will have during this study, through a satisfaction questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Age between 5 and 55 years
* Any level of GMFCS (Gross Motor Function Classification System)
* The patient consent to participate in the study
* Diagnosis of spastic cerebral palsy
* Triceps Surae spasticity in them.
* The dynamic foot deformity.
* Extensibility between 0 ° and 20 ° in dorsal flexion passive way.
* Do not be diagnosed important cutaneous alterations.

Exclusion Criteria:

* Associate neuromuscular disease.
* Surgical Intervention to augment the balance articulate and / or reduce the spasticity in the last six months.
* Fixed foot deformity.
* Etiology of factors:

or genetic bone disorders / disturbances soft parts. Position with anomalies or alterations in soft parts or bone alterations (mechanical).

* Unable to follow the treatment.
* Allergy to botulinum toxin.

Ages: 5 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2014-09; Primary Completion 2015-06 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
muscle elongation of spastic muscle will be evaluated using composite measure of muscular extensibility and their traction reflex with goniometry | up to three months

SECONDARY OUTCOMES:
Evaluate the patients perceive pain | after each therapy
  It shall be assessed by visual analog scale
Ascertain if the type of GMFCS has an influence on the improvement of these two treatments. Qualitative registation to achieve the percepcion and experience that have made the treatment received the patient/family. | at the end to study
To undergo a qualitative registration to know the perception and experience that patient/family will have during this study | at the end to study

CONTACTS AND LOCATIONS:
Overall Officials: Vidal Novellas, Principal Investigator — Aspace. Association of Cerebral Palsy
Locations (1):
- Centro Piloto Arcangel Sant Gabriel. ASPACE, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes